CLINICAL TRIAL: NCT02984020
Title: Korean Post-marketing Surveillance for Xeljanz(Registered) in Rheumatoid Arthritis and Psoriatic Arthritis Patients
Brief Title: Korean Post-marketing Surveillance for Xeljanz
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921249
Record Dates: First submitted 2016-11-03; First posted 2016-12-06 (Estimated); Results first posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this study is to identify any problems and questions with respect to the safety and efficacy of Xeljanz during the post-marketing period as required by the regulation of MFDS.

ELIGIBILITY:
Inclusion Criteria:

To be included in the study all patients will have received at least 1 dose of Xeljanz for the treatment of the following indication as per local labelling. Moderately to severely active RA in adult patients who have had an inadequate response or intolerance to previous therapy with at least 1 biological DMARD. Or Active psoriatic arthritis (PsA) who have had an inadequate response or intolerance to previous antirheumatic drugs (DMARDs)

Exclusion Criteria:

1. Patients with a history of hypersensitivity to any ingredients of the product.
2. Patients with serious infection (eg, sepsis) or active infection including localized infection.
3. Patients with active tuberculosis.
4. Patients with severe hepatic function disorder.
5. Patients with an absolute neutrophil count (ANC) <500 cells/mm3.
6. Patients with a lymphocyte count <500 cells/mm3.
7. Patients with a hemoglobin concentration <8 g/dL.
8. Pregnant or possibly pregnant women.
9. Because of lactose contained in this drug, it should not be administered to patients with hereditary problems of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.

According to Contraindication on label, the investigator should discontinue the patient's treatment if the laboratory test results are as below Patients with an absolute neutrophil count (ANC) <500 cells/mm3 Patients with a hemoglobin level <8 g/dL

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult rheumatoid arthritis or psoriatic arthritis taking tofacitinib within label as Ministry of Food and Drung Safety in Korea has approved
Sampling Method: Non-Probability Sample
Enrollment: 1041 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (49):
- South Korea (49):
  - Soonchunhyang University Cheonan Hospital, Department of Rheumatology, Chunan-si, Chungcheongnam-do
  - Keimyung University Dongsan Medical Center, Jung-Gu, Daegu
  - Kongyang University Hospital / Rheumatology, Seogu, Daejon
  - Myongji Hospital / Rheumatology, Goyang-si, Deogyang-gu
  - Kyung Hee University Hospital at Gangdong / Rheumatology, Seoul, Gangdong-gu
  - VHS Medical Center / Rheumatologist, Seoul, Gangdong-gu
  - Hallym University Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do
  - Chosun University Hospital, Rheumatism Department, Donggu, Gwang JU
  - Division of Rheumatology, Seongnam-si, Gyeongg-do
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Yangsan Hospital-Pusan National University, Yangsan, Gyeongsangnam-do
  - Chonbuk National University Hospital, Department of Rheumatology, Jeonju, Jeollabuk-do
  - Wonkwang University Hospital / Division of Rheumatology, Iksan, Jeonlabuk-do
  - Ajou University Hospital, Department of Rheumatology, Suwon, Kyeongki-do
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Inje University Busan Paik hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Inje University Haeundae Paik Hospital, Busan
  - Chungbuk National University Hospital, Chungcheongbuk-do
  - Daegu Catholic University Medical Center, Department of Rheumatology, Daegu
  - Eulji University Hospital, Internal Medicine, Rheumatology, Daejeon
  - Yongin Severance Hospital, Giheung-gu, Yongin-si, Gyeonggi-do
  - Inje University IlsanPaik Hospital, Goyang-si, Gyeonggi-do
  - Dongguk University Ilsan Medical Center, Gyeonggi-do
  - Gachon University Gil Hospital, Incheon
  - Division of Rheumatology, Incheon
  - Jeju National University Hospital, Jeju Special Self-Goverming Province
  - Division of Rheumatology, Metropolitan City, Daejeon
  - Pusan National University Hospital, Pusan
  - Dong-A University Hospital, Pusan
  - Hanyang Rheuma Uhm Wan-Sik Clinic, Seoul
  - Division of Rheumatology, SMG-SNU Boramae Medical Center, Seoul
  - Seoul National University Hospital, Department of Internal Medicine, Seoul
  - Seoul National University Hospital, Rheumatology, Internal Medicine, Seoul
  - Kyung Hee University Hospital, Seoul
  - Hanyang University Hospital, Department of Rheumatology, Seoul
  - Kyunghee University East-West Neo Medical Center, 149 Sangil-dong, Gangdong-gu, Seoul
  - Samsung Medical Center, Division of Rheumatology, Department of Medicine, Seoul
  - The Catholic University of Korea, Kangnam St. Mary's Hospital/ Rheumatology, Internal Medicine, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital/ Rheumatology, Internal Medicine, Seoul
  - Eulji Medical Center, Seoul
  - Soonchunhyang University Hospital Seoul/Department of Rheumatology, Seoul
  - Konkuk University Medical Center, Seoul
  - Division of Rheumatology, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a study conducted in Korea. The investigator enrolled participants to whom Xeljanz was prescribed for the first time according to the local product document and who agreed to participate in this study. Xeljanz was administered according to the "Dosage and Administration" of the approved labeling.
  Xeljanz was medicated by the investigator's prescription under usual clinical practice.
Groups:
- Post-Marketing Surveillance: Xeljanz: Participants with moderately to severely active rheumatoid arthritis (RA) who had an inadequate response or intolerance to methotrexate were observed during this post-marketing surveillance (PMS) study. The entire study period was approximately 6 years.
Period: Overall Study
Arm/Group | Post-Marketing Surveillance: Xeljanz
Started | 1041
Completed | 1009
Not Completed | 32
Not completed — Experienced off-label use against Xeljanz local product document | 21
Not completed — Not met the inclusion/exclusion criterion | 9
Not completed — Other significant protocol violation | 2

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who received at least 1 dose of Xeljanz according to local product document and was assessed for safety information.
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 1009
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Mean | 55.04 (12.64)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 126
  >= 40 years and < 50 years | 195
  >= 50 years and < 60 years | 305
  >= 60 years and < 70 years | 258
  >= 70 years | 125
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 852
  Male | 157
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Indication, RA/PsA [Count of Participants; unit: Participants] — RA = rheumatoid arthritis, PsA = psoriatic arthritis.
  Participants
    RA | 1009
    PsA | 0
Duration of the disease, Continuous [Mean (Standard Deviation); unit: Months] — The duration of disease since the date that the participant was initially diagnosed with RA or PsA was recorded.
  Months | 98.36 (80.77)
Duration of the disease, Customized [Count of Participants; unit: Participants] — The duration of disease since the date that the participant was initially diagnosed with RA or PsA was recorded.
  Participants
    < 3 years | 219
    >= 3 years and < 6 years | 193
    >= 6 years and < 9 years | 146
    >= 9 years and < 12 years | 121
    >= 12 years | 214
    Unknown | 116
Severity of disease activity, High/Moderate/Low/Not assessed [Count of Participants; unit: Participants] — Disease Activity Score 18 (DAS28) >5.1 is considered to be indicative of high disease activity; DAS28 >3.2 and ≤5.1 indicates moderate disease activity; DAS28 ≤3.2 indicates low disease activity.
  Participants
    High (DAS28 > 5.1) | 874
    Moderate (DAS28 > 3.2 and <= 5.1) | 135
    Low (DAS28 <= 3.2) | 0
    Not assessed | 0
Radiologic progression, Yes/No/Not assessed [Count of Participants; unit: Participants] — Radiologic progression based on clinically relevant evaluation methods, such as X-ray, ultrasonography, or magnetic resonance imaging was recorded.
  Participants
    Yes | 506
    No | 290
    Not assessed | 213
Status of latent tuberculosis, Yes/No/Unknown [Count of Participants; unit: Participants]
  Yes | 226
  No | 770
  Unknown | 13
Herpes zoster Vaccination, Yes/No/Unknown [Count of Participants; unit: Participants]
  Yes | 115
  No | 407
  Unknown | 487
Smoking, Ex-smoking/Current smoking/Non-smoking/Unknown [Count of Participants; unit: Participants]
  Ex-smoking | 64
  Current smoking | 57
  Non-smoking | 706
  Unknown | 182
Renal disorder, Yes/No [Count of Participants; unit: Participants]
  Yes | 19
  No | 990
Hepatic disorder, Yes/No [Count of Participants; unit: Participants]
  Yes | 40
  No | 969
Allergic history, Yes/No [Count of Participants; unit: Participants]
  Yes | 25
  No | 984
Prior rheumatoid arthritis therapy, Yes/No [Count of Participants; unit: Participants]
  Yes | 890
  No | 119
Concomitant medication, Yes/No [Count of Participants; unit: Participants] — Number of participants who received concomitant medication were recorded.
  Participants
    Yes | 997
    No | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs), Adverse Drug Reactions (ADRs), Serious Adverse Events (SAEs) and Serious Adverse Drug Reactions (SADRs)
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. SAE was any untoward medical occurrence that at any dose resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; congenital anomaly/birth defect. An ADR was any untoward medical occurrence attributed to Xeljanz in a participant who received Xeljanz. SADR was an ADR resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience; initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly/birth defect. Relatedness to Xeljanz was assessed by the physician.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: The safety analysis set included all participants who had received at least 1 dose of Xeljanz according to local product document and had been assessed for safety information including AEs by investigator.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 1009
Participants
  Adverse Events(AEs) | 261
  Adverse Drug Reactions(ADRs) | 148
  Serious Adverse Events(SAEs) | 40
  Serious Adverse Drug Reactions(SADRs) | 20
  Adverse Events of Special Interest | 21
  Adverse Drug Reactions of Special Interest | 16

2. Primary Outcome: Number of Participants With Unexpected AEs, Unexpected SAEs, Unexpected ADRs and Unexpected SADRs
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. SAE was any untoward medical occurrence that at any dose resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity; congenital anomaly/birth defect. An ADR was any untoward medical occurrence attributed to Xeljanz in a participant who received Xeljanz. SADR was any SAE that is attributed to Xeljanz. Relatedness to Xeljanz was assessed by the physician. An unexpected AE was an AE with a difference in nature, severity, specificity, or outcome, compared to the product licensure/safety notification of the drug. Unexpected ADRs were unexpected AEs that were, in the investigator's opinion, of causal relationship to the study treatment.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 1009
Participants
  Unexpected Adverse Events | 99
  Unexpected Adverse Drug Reactions | 31
  Unexpected Serious Adverse Events | 11
  Unexpected Serious Adverse Drug Reactions | 1

3. Primary Outcome: Duration of Adverse Events
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. Only participants with available data are reported.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 163
Days | 26 [0 to 320]

4. Primary Outcome: Number of Participants With Adverse Events by Their Severity
Description: The evaluation of AE severity was done according to the following categories: mild: not causing any significant problem to the participant. Administration of medicinal product continues without dose adjustment. Moderate: causes a problem that dose not interfere significantly with usual activities or the clinical status. Dose of the medical product is adjusted or other therapy is added due to the AE. Severe: causes a problem that interferes significantly with usual activities or the clinical status. The medicinal product is stopped due to the AE. Only participants with available severity assessment data are reported.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 261
Participants
  Mild | 201
  Moderate | 82
  Severe | 7

5. Primary Outcome: Number of Participants With Adverse Events by Their Outcome
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. The outcomes of AE included recovered, recovered with sequelae, recovering, not recovered and unknown. One participant may experience more than one event hence one participant may be included in more than one category specified below. Only participants with available outcome assessment are reported.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 261
Participants
  Recovered | 200
  Recovered with sequelae | 1
  Recovering | 43
  Not recovered | 38
  Unknown | 7

6. Primary Outcome: Number of Participants With Adverse Events by Their Seriousness Criteria
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. The seriousness criteria for AEs included results in death, is life-threatening, requires inpatient hospitalization or prolongation of hospitalization, results in persistent or significant disability/incapacity, results in congenital anomaly/birth defect, other important medical event. Only participants with available seriousness assessment data are reported.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 261
Participants
  Results in death | 2
  Is life-threatening | 1
  Requires inpatient hospitalization or prolongation of hospitalization | 40
  Results in persistent or significant disability/incapacity | 0
  Results in congenital anomaly/birth defect | 0
  Is an important medical event | 0
  Non-SAE | 238

7. Primary Outcome: Number of Participants With Adverse Events by Their Action Taken With Regard to Xeljanz
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship. The action taken with regard to the medicinal product included: permanently discontinued, temporarily discontinued or delayed, dose reduced, dose increased, no change, not applicable. Only participants with available action taken assessment data are reported.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 261
Participants
  Permanently discontinued | 45
  Temporarily discontinued or delayed | 35
  Dose reduced | 14
  No change | 188
  Not applicable | 4

8. Primary Outcome: Number of Participants With Adverse Events by Their Causality to Xeljanz
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship. The causality of AEs to Xeljanz were assessed by physician according to the following criteria: certain, probable/likely, possible, unlikely, conditional/unclassified and unassessible/unclassifiable. One participant may experience more than one event hence, one participant may be included in more than one category specified below. Only participants with available causality assessment data are reported.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 261
Participants
  Certain | 1
  Probable/likely | 9
  Possible | 101
  Unlikely | 134
  Conditional/unclassified | 17
  Unaccessible/unclassifiable | 25

9. Primary Outcome: Number of Participants With Adverse Events According to Demographic Characteristics
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. Number of participants with AEs classified according to the following demographic characteristics: sex: male and female; age: less than (<) 40 years, greater than or equal to (>=) 40 and < 50 years and >= 50 years and <60 years; >= 60 and <70 years; geriatric (>=65 years). Only participants with available demographic and AE assessment data are reported.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 261
Participants
  Sex: Male | 36
  Sex: Female | 225
  Age: < 40 years | 35
  Age: >= 40 years and < 50 years | 48
  Age: >= 50 years and < 60 years | 79
  Age: >= 60 years and < 70 years | 63
  Age: >= 70 years | 36
  Geriatric (>= 65 years) | 67

10. Primary Outcome: Number of Participants With Adverse Events According to Other Baseline Characteristics
Description: Other baseline characteristics included: indication; duration of the disease; severity of disease; radiologic progression; status of latent tuberculosis; herpes zoster vaccination; smoking; prior rheumatoid arthritis therapy; medical history; renal disorder; hepatic disorder; allergic history; concomitant medication; duration of administration. Only participants with available other baseline characteristics and AE assessment data are reported.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 261
Participants
  Indication: RA | 261
  Indication: PsA | 0
  Duration of the disease: < 3 years | 55
  Duration of the disease: >= 3 years and < 6 years | 47
  Duration of the disease: >= 6 years and < 9 years | 25
  Duration of the disease: >= 9 years and < 12 years | 35
  Duration of the disease: >= 12 years | 70
  Duration of the disease: Unknown | 29
  Severity of disease activity: High (DAS28 > 5.1) | 226
  Severity of disease activity: Moderate (DAS28 > 3.2 and <= 5.1) | 35
  Severity of disease activity: Low (DAS28 <= 3.2) | 0
  Severity of disease activity: Not assessed | 0
  Radiologic progression: Yes | 132
  Radiologic progression: No | 62
  Radiologic progression: Not assessed | 67
  Status of latent tuberculosis: Yes | 52
  Status of latent tuberculosis: No | 206
  Status of latent tuberculosis: Unknown | 3
  Herpes zoster Vaccination: Yes | 33
  Herpes zoster Vaccination: No | 125
  Herpes zoster Vaccination: Unknown | 103
  Smoking: Ex-smoking | 18
  Smoking: Current smoking | 16
  Smoking: Non-smoking | 188
  Smoking: Unknown | 39
  Prior rheumatoid arthritis therapy: Yes | 238
  Prior rheumatoid arthritis therapy: No | 23
  Medical history: Yes | 209
  Medical history: No | 52
  Renal disorder: Yes | 6
  Renal disorder: No | 255
  Hepatic disorder: Yes | 13
  Hepatic disorder: No | 248
  Allergic history: Yes | 11
  Allergic history: No | 250
  Concomitant medication: Yes | 259
  Concomitant medication: No | 2
  Duration of administration: < 6 months | 75
  Duration of administration: >= 6 months and < 7 months | 135
  Duration of administration: >= 7 months | 39
  Duration of administration: Unknown | 12

11. Primary Outcome: Number of Participants With Adverse Events - Multivariate Logistic Regression Analysis
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. Logistic regression analysis of multivariate analysis was performed and presented an odds ratio with 95% confidence interval to identify the factors that affect occurrence of AEs in demography and baseline characteristics, or concomitant treatment status, etc.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 1009
Participants | 261
Statistical Analysis 1: Comparison: Post-Marketing Surveillance: Xeljanz; Test type: Other; p < 0.0001, Regression, Logistic; Multiple logistic regression including total treatment duration of Xeljanz as factor; Odds Ratio (OR) = 0.77, 95% CI [0.69 to 0.86]
Statistical Analysis 2: Comparison: Post-Marketing Surveillance: Xeljanz; Test type: Other; p < 0.0001, Regression, Logistic; Multiple logistic regression including other past/present disease as factor; Odds Ratio (OR) = 2.43, 95% CI [1.64 to 3.59]

12. Primary Outcome: Number of Geriatric Participants With Adverse Events and Adverse Drug Reactions
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. An ADR was any untoward medical occurrence attributed to Xeljanz in a participant who received Xeljanz.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: The population included geriatric participants (aged >=65 years) in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 238
Participants
  Adverse Events | 67
  Adverse Drug Reactions | 43

13. Primary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions - Renal Disorder
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. An ADR was any untoward medical occurrence attributed to Xeljanz in a participant who received Xeljanz. Renal disorder was judged by the investigator.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: The population included participants with renal disorder in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 19
Participants
  Adverse Events | 6
  Adverse Drug Reactions | 5

14. Primary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions - Hepatic Disorder
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. An ADR was any untoward medical occurrence attributed to Xeljanz in a participant who received Xeljanz. Hepatic disorder was judged by the investigator.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: The population included participants with hepatic disorder in the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 40
Participants
  Adverse Events | 13
  Adverse Drug Reactions | 7

15. Primary Outcome: Number of Participants With Adverse Events and Adverse Drug Reactions - Other Than Safety Analysis Population
Description: An AE was any untoward medical occurrence in a participant administered a medicinal or nutritional product (including pediatric formulas) without regard to possibility of a causal relationship with product treatment or usage. An ADR was any untoward medical occurrence attributed to Xeljanz in a participant who received Xeljanz. AEs and ADRs for participants excluded from the safety analysis population were reported. The reason for exclusion included: not met the inclusion criteria/met exclusion criteria; off-label use; other significant protocol violation.
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years)
Population: The population included participants excluded from the safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 31
Participants
  Adverse Events | 14
  Adverse Drug Reactions | 9

16. Secondary Outcome: Change From Baseline in DAS28 (ESR)
Description: DAS28 is a modified version of the original Disease Activity Score (DAS). It is a quantitative measure of disease activity used to monitor the treatment or RA. DAS28 (erythrocyte sedimentation rate [ESR]) was calculated from: DAS28 (ESR) = 0.56*√(tender joint counter [TJC] 28) + 0.28*√(swollen joint count [SJC] 28) + 0.014*VAS+ 0.70*ln(ESR), where VAS = visual analogue scale. Total score range: 0-9.4, higher score=more disease activity.
Time Frame: From Baseline to 6 months after treatment (through study completion, up to approximately 6 years)
Population: The analysis set included all participants who received at least 1 dose of Xeljanz and were available for an effectiveness assessment.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 841
Scores on a scale | -2.35 (1.11)

17. Secondary Outcome: Change From Baseline in DAS28 (CRP)
Description: DAS28 is a modified version of the original Disease Activity Score (DAS). It is a quantitative measure of disease activity used to monitor the treatment or RA. DAS28-3 ( C-reactive protein [CRP]) was calculated from the swollen joint count (SJC) and tender joint count (TJC) using the 28 joints count and CRP (mg/L). Total score range: 0 to 9.4, higher score indicated more disease activity.
Time Frame: From Baseline to 6 months after treatment (through study completion, up to approximately 6 years)
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 455
Scores on a scale | -2.42 (1.10)

18. Secondary Outcome: Number of Participants With EULAR Response
Description: European League Against Rheumatism (EULAR) response is a DAS-based response criteria that classifies individual participants as none, moderate, or good responders, depending on the extent of change and the level of disease activity reached. Participants with improvement in DAS28 from baseline >1.2 and DAS28 based EULAR <=3.2 were good responders; participants with improvement in DAS28 from baseline >0.6 and <=1.2 and DAS28 based EULAR >3.2 and <=5.1 were moderate responders; participants with improvement in DAS28 from baseline <=0.6 and DAS28-based EULAR >5.1 were none responders.
Time Frame: From Baseline to 6 months after treatment (through study completion, up to approximately 6 years)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 903
Participants
  Good | 404
  Moderate | 446
  None | 53

19. Secondary Outcome: Number of Participants With an American College of Rheumatology 20% (ACR20) Response at Month 6
Description: ACR20 response: ≥20% improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and CRP.
Time Frame: From Baseline to 6 months after treatment (through study completion, up to approximately 6 years)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 903
Participants | 209

20. Secondary Outcome: Number of Participants With Effectiveness
Description: The variables included DAS28, EULAR response, and ACR20 response. The investigator made the assessment of the overall effectiveness as improved, no change, or aggravated, based on each test results and clinical judgment. No change and aggravated were classified as ineffective.
Time Frame: From Baseline to 6 months after treatment (through study completion, up to approximately 6 years)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 903
Participants
  Effective: Improved | 853
  Ineffective: No change | 36
  Ineffective: Aggravated | 14

21. Secondary Outcome: Number of Participants With Effectiveness by Demographic Characteristics
Description: The variables included DAS28, EULAR response, and ACR20 response. The investigator made the assessment of the overall effectiveness as improved, no change, or aggravated, based on each test results and clinical judgment.
Time Frame: From Baseline to 6 months after treatment (through study completion, up to approximately 6 years)
Population: The analysis set included all participants who received at least 1 dose of Xeljanz and were available for an effectiveness assessment and with improved effectiveness.
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 853
Participants
  Sex: Male | 128
  Sex: Female | 725
  Age: < 40 years | 110
  Age: >= 40 years and < 50 years | 162
  Age: >= 50 years and < 60 years | 256
  Age: >= 60 years and < 70 years | 219
  Age: >= 70 years | 106
  Geriatric (>= 65 years) | 200

22. Secondary Outcome: Number of Participants With Improved Effectiveness - Multivariate Logistic Regression Analysis
Description: The variables included DAS28, EULAR response, and ACR20 response. The investigator made the assessment of the overall effectiveness as improved, no change, or aggravated, based on each test results and clinical judgment. Logistic regression analysis of multivariate analysis was performed and presented as odds ratios with 95% confidence interval to identify the factors that affected classified overall assessment (effective/ineffective) in demography and baseline characteristics of the participants.
Time Frame: From Baseline to 6 months after treatment (through study completion, up to approximately 6 years)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Post-Marketing Surveillance: Xeljanz
Number analyzed (Participants) | 903
Participants | 853
Statistical Analysis 1: Comparison: Post-Marketing Surveillance: Xeljanz; Test type: Other; p = 0.0053, Regression, Logistic; Multiple logistic regression including total duration of treatment with Xeljanz as factor; Odds Ratio (OR) = 1.42, 95% CI 2-sided [1.11 to 1.82]

ADVERSE EVENTS:
Time Frame: From first dose for Xeljanz to 28 days after last dose (through study completion, up to approximately 6 years).
Arm/Group | Post-Marketing Surveillance: Xeljanz
All-Cause Mortality (participants affected / at risk) | 2/1009
Serious Adverse Events (participants affected / at risk) | 40/1009
Other Adverse Events (participants affected / at risk) | 261/1009
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Post-Marketing Surveillance: Xeljanz (N=1009)
Cardiac failure congestive (Cardiac disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 5
Influenza (Infections and infestations) | 2
Peritonsillar abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pyelonephritis acute (Infections and infestations) | 2
Sinusitis fungal (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral infarction (Nervous system disorders) | 1
Mononeuritis (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Post-Marketing Surveillance: Xeljanz (N=1009)
Anaemia (Blood and lymphatic system disorders) | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Tachycardia (Cardiac disorders) | 1
Type IIa hyperlipidaemia (Congenital, familial and genetic disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 2
Diplopia (Eye disorders) | 1
Dry eye (Eye disorders) | 2
Eye pain (Eye disorders) | 2
Vision blurred (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 3
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 7
Enteritis (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastritis erosive (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 9
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 3
Chills (General disorders) | 1
Face oedema (General disorders) | 8
Fatigue (General disorders) | 2
Generalised oedema (General disorders) | 2
Oedema peripheral (General disorders) | 7
Swelling face (General disorders) | 3
Gallbladder polyp (Hepatobiliary disorders) | 1
Hepatic steatosis (Hepatobiliary disorders) | 2
Liver disorder (Hepatobiliary disorders) | 1
Abscess limb (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Cystitis (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 23
Influenza (Infections and infestations) | 3
Nasopharyngitis (Infections and infestations) | 31
Oral herpes (Infections and infestations) | 2
Periodontitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Pyelonephritis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Tinea cruris (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 1
Vaginal infection (Infections and infestations) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase abnormal (Investigations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase abnormal (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood cholesterol increased (Investigations) | 1
Blood pressure increased (Investigations) | 2
Hepatic enzyme increased (Investigations) | 1
High density lipoprotein increased (Investigations) | 5
Liver function test abnormal (Investigations) | 2
Liver function test increased (Investigations) | 1
Weight decreased (Investigations) | 2
Weight increased (Investigations) | 2
Dyslipidaemia (Metabolism and nutrition disorders) | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Cerebral artery occlusion (Nervous system disorders) | 1
Cerebral artery stenosis (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 13
Headache (Nervous system disorders) | 6
Hypoaesthesia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Dysuria (Renal and urinary disorders) | 3
Renal cyst (Renal and urinary disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Breast pain (Reproductive system and breast disorders) | 1
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1
Scrotal pain (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 3
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 5
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclosure previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-04-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT02984020/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/20/NCT02984020/SAP_001.pdf